CLINICAL TRIAL: NCT00813579
Title: Study of Prospective Assessment of Living Kidney Donors:Pre and Post Donation
Brief Title: Study of Prospective Assessment of Living Kidney Donors: Pre and Post Donation
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Mansoura University (Other)
Responsible Party: Ayman Maher Nagib Kerilos, Mansoura U
Other Study IDs: 1212
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-12

CONDITIONS: Kidney Donation
Keywords: assess the safety of living kidney donation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a prospective assessment of 80 living kidney donors.

ELIGIBILITY:
Inclusion Criteria:

* Donors are suitable candidate for living donation
* Male or female donors minimum 21 years maximum 65 years of age
* Donors has been fully informed and has given written informed consent

Exclusion Criteria:

* Donors has diabetes mellitus or hypertension.
* Donors is pregnant or breastfeeding.
* Donors is known to be HCV,HBV,HIV positive or has significant liver disease.
* Donors with malignancy or history of malignancy.
* Donors has systemic or localized major infection.
* Donors is participating or has participated in another clinical trial.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prspective one arm study of 80 live kidney donors . Pre and post donation evaluation(clinical evaluation BLOOD PRESURE BMI, Laboratory evaluaion of renal hepatic functions ,lipid profil, blood sugar, complet blood count,urinanalysis for protein creatinine ratio ,psychological assesment and renal ultrasound for kidney size and any abnormality at 3,6,12,24 months post donation.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-01 (Estimated); Study Completion 2011-01 (Estimated)

REFERENCES:
- [Derived] Nagib AM, Refaie AF, Hendy YA, Elfawal MA, Shokeir AA, Bakr MA, Neamattala AH, Hamdy AF, Mahmoud KM, Ismail AM, Ghoneim MA. Long term prospective assessment of living kidney donors: single center experience. ISRN Nephrol. 2014 Jan 23;2014:502414. doi: 10.1155/2014/502414. eCollection 2014. PMID 24967244